CLINICAL TRIAL: NCT05664542
Title: Efficacy of Erector Spinae Block With Ropivacaine and Dexmedetomidine on Opioid Consumption After Lumar Spine Surgeries - A Randomised Controlled Trial
Brief Title: Erector Spinae Block With Ropivacaine and Dexmedetomidine on Opioid Consumption After Lumar Spine Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Principal investigator, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SFH-ESPB Dex
Record Dates: First submitted 2022-11-20; First posted 2022-12-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: 2 groups, one with block and other with no block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Procedure will be done after patient will undergo GA for surgery. Medications will be prepared by anesthetist not involved in the study. The nurse/doctor who will assess the outcome will not know the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB group (Experimental): this group will receive ESPB using ropivacaine and dexmedetomidine
  Interventions: Other: ESPB (regional Block); Drug: ropivacaine and dexmedetomidine
- Control group (No Intervention): this group will not receive any block

INTERVENTIONS:
Other: ESPB (regional Block) — ESPB is regional block in which we will use 0.2 % ropivacaine and dexmedetomidine
  Arms: ESPB group
Drug: ropivacaine and dexmedetomidine — 0.2 % ropivacaine and dexmedetomidine
  Arms: ESPB group

SUMMARY:
The aim of this study is to investigate the role of 0.5 micrograms/kg of dexmedetomidine with 0.2 % ropivacaine in erector spinae block in reducing opioid consumption for patients undergoing lumbar spine surgeries. This study will help in understanding the role of adding dexmdetomidine to ropivacaine in erector spinae block in reducing opioid consumption after lumbar spine surgeries

DETAILED DESCRIPTION:
A number of adjuvants have been used with local anesthetics including dexamethasone, nalbuphine and dexmedetomidine etc with the aim of improving quality and duration of peripheral nerve blocks. Dexmedetomidine is a potent alpha-2 agonist which can prolong the duration of regional anesthesia block when used in combination with local anesthetics. Although, there is no consensus on the dose of dexmedetomidine for peripheral nerve block considering the fact that it can lower heart rate and blood pressure intraoperatively. Investigators therefore, planned this randomised controlled trial to investigate the role of 0.5 micrograms/kg of dexmedetomidine with 0.2 % ropivacaine in erector spinae block for patients undergoing lumbar spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years, scheduled to undergo lumbar spine surgeries with an ASA score of 1 to 3 will be included in the study

Exclusion Criteria:

* Patients who refused enrollment or later requested removal for the study, those who are unable to give informed consent and patients with either contraindications for regional anesthesia, known allergy to local anesthetics or dexmedetomidine, bleeding diathesis, use of anticoagulants or corticosteroids, inability to operate patient controlled analgesia (PCA) system, psychiatric disorders or use of psychiatric medications will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
24 hours opioid consumption | 24 hours
  opioid consumption in mg during first 4 hours postoperatively

SECONDARY OUTCOMES:
pain score | 24 hours
  pain score in Numerical rating score during first 24 hours postoperatively
Occurrence of postoperative nausea and vomiting (PONV) | 24 hours
  Occurrence of postoperative nausea and vomiting (PONV) during first 24 hours
Occurrence of drowsiness | 24 hours
  Occurrence of drowsiness in 24 hours will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Anwar ul Huda, FRCA, Principal Investigator — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF